CLINICAL TRIAL: NCT05542888
Title: Effects of Antenatal Exercises With Sacroiliac Joint Mobilization in Pregnancy Related Pelvic Girdle Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/16
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy Related Pelvic Girdle Pain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial which will consist of two groups. Once will recieve conventional physcial therapy and the sencond will recieve conventional physcial therapy with sacroiliac joint mobilization.Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a another person who will be unaware of the group the particpant belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Postural education Hot pack(10 min) Antenatal exercises(i.e. deep breathing(5 min), stretching(5 min), kegel exercises(5 min), Mitchells physiologic relaxation technique(10 min) and walk(10 min) Sacro iliac joint mobilization(5 min) Total duration:50 min/session
  Interventions: Procedure: Sacroiliac joint mobilization; Procedure: Standard therapy
- Control group (Active Comparator): Postural education Hot pack(10 min) Antenatal exercises(i.e.deep breathing(5 min), stretching(5 min), kegel exercises(5 min), Mitchells physiologic relaxation technique(10 min) and walk(10 min) Total duration:45 min/session
  Interventions: Procedure: Standard therapy

INTERVENTIONS:
Procedure: Sacroiliac joint mobilization — Sacroiliac joint mobilization will be performed with the patient in side lying position in which grade I,II pain relief mobilization will be given in PA direction.It will be given as 1 set of 30 oscillations per session, 3 times per week for 4 weeks.
  Arms: Experimental group
Procedure: Standard therapy — Postural education, Hot pack, Antenatal exercises

SUMMARY:
Pelvic girdle pain is the frequently occuring pregnancy-related musculoskeletal condition.It is defined as the pain experienced between the posterior iliac crest and the gluteal region, particularly in the sacroiliac joint.This condition is associated with difficulties in activities of daily life such as standing, walking, working and sleeping hence affecting the quality of life.Various management strategies including antenatal exercises, sacro iliac joint belt, kinesiotaping, sacro iliac joint mobilization etc are used for treating the pelvic girdle pain.Different studies have shown the positive results of antenatal exercises, sacro iliac joint belt and kinesiotaping on the pelvic girdle pain but there is lack of data available to establish the efficacy of sacro iliac joint mobilization on pregnancy-related pelvic girdle pain.So this study aims tofulfill this gap by comparing the effects of antenatal exercises with sacro iliac jpint mobilization on pelvic pain, function and disability in pregnancy-related pelvic girdle pain

DETAILED DESCRIPTION:
Pelvic girdle pain is defined as the pain experienced between the posterior iliac crest and the gluteal region, particularly in the sacro iliac joint.It is characterized by pain, instability, limitations in mobility and functioning of the pelvic region.This condition is found to be associated with difficulties in activities of daily life such as standing, walking, working and sleeping hence, affecting the quality of life.Pelvic girdle pain is on of the major preganacy-related problems that affects about 50% of the pregnant females.Previous studies have shown that about 33-50% of the women repost pelvic girdle pain before 20 weeks of gestation and the the prevalavce may reach 60-70% in late pregnancy.Different management strategies including antenatal exercises, sacro iliac joint belt, kinesiotaping, sacro iliac joint mobilization etc are used to treat pelvic girdle pain.Different studies have shown the positive results of antenatal exercises, sacro iliac joint belt and kinesiotaping but there is dearth of evidence to establish the efficacy of sacro iliac joint mobilization on pregnancy-related pelvic girdle pain.This study aims to fulfill this gap by comparing the effects of antenatal exercises with sacro iliac joint mobilization on pelvic pain, function and disability.

This randomized control trial will be conducted in Obs&Gynae Opd of Fauji Foundation Hospital using non-probability purposive sampling.Participants will be briefed regarding the study objectives, procedure, risks and benefits of treament, voluntary participation and right to withdraw.Written informed consent will be taken from all the participants before conducting the research.Details of exercise program will be explained to them.Screening will be done by using PAR Q.Dignostic tests will be applied to confirm the pelvic girdle pain.FABERs test and Posterior Pelvic Pain Provocation test will be used for this purpose.Then the selected participants will be randomized into 2 groups(experimental group and control group)via lottery method. Participants will complete Numeric Rating Pain Scale(NRPS) for pain, Pelvic Girdle Questionnaire for disability measurement and will perform Active Straight Leg raise test(ASLR) to measure pelvic function.All of these measurements will be taken at baseline, after 2 weeks and then after 4 weeks of intervention.

The treatment protocol of both groups is as follows:

Group 1(Control group):Postural education, hot pack, antenatal exercises(i.e deep breathing, stretching, kegel exercises, Mitchells physiologic relaxation technique and walk.

Group 2(Experimental group):Postural ecucation, hot pack, antenatal exercises(i.e deep breathing, stretching, kegel exercises, Mitchells physiologic relaxation technique and walk) and sacro iliac joint mobilization in side lying position(1 set of 30 oscillatios per session)

ELIGIBILITY:
Inclusion Criteria:

* Both primiparous and multiparous gestational women of age 18-40 years
* Gestational age: 13-24 weeks of 2nd trimester

Exclusion Criteria:

-History of: Miscarriages Early Neonatal Deaths Intra-uterine growth retardation Premature rupture of membranes Arthritis Twins/triplets pregnancies

* Present complain of Pregnancy Induced Hypertension(HIP)
* Placenta previa

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 32 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain intensity will be measured on numeric rating pain scale. It consists of 11 points( interval 0-10), where 0 corresponds to no pain and 10 corresponds to worst pain imaginable. A graphical representation of 11 spaces is used for patients own evaluation of his or her pain.
Disability | 4 weeks
  The Pelvic Girdle Questionnaire(PGQ) is a condition-specific tool that assesses activity limitation and symptoms in patients with pelvic girdle pain .It consists of 20 activity items and 5 symptoms items scored on a 4-point response scale .Each question is scored from "Not at all" to "to a large extent". Items scores are summed and transformed to yield a score of 0 to 100, where 100 is the worst possible score
Pelvic function | 4 weeks
  The Active Straight Leg Raise Test is a functional test used to assess pelvic girdle pain. It consists of a 6-point scale: not difficult at all=0, minimally difficult=1, somewhat difficult=2, fairly difficult=3, very difficult=4, unable to do=5. The scores of both sides are added so that the summed score can range from 0-10. Impairment is considered severe if the summed bilateral score is at least 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan